CLINICAL TRIAL: NCT06884696
Title: Study of Placental Inflammation in Gestational Diabetes: the Role of the Inflammosome NLRP3 and the Scavenger Receptor of Inflammatory Chemokines D6
Brief Title: Study of Placental Inflammation in Gestational Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 4978
Record Dates: First submitted 2025-03-05; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-06

CONDITIONS: Gestational Diabetes Mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Specimen Collection; Placental Extracts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with gestational diabetes mellitus (Experimental): Blood and placenta sampling will be obtained from cases= women with gestational diabetes mellitus
  Interventions: Other: Blood samples for inflammatory markers; Other: Placental Extract
- Healthy women with uncomplicated pregnancy (Experimental): Blood and placenta sampling will be obtained from controls= women with uncomplicated pregnancy
  Interventions: Other: Blood samples for inflammatory markers; Other: Placental Extract

INTERVENTIONS:
Other: Blood samples for inflammatory markers — Blood sampling
Other: Placental Extract — Placental sampling after caesarean section

SUMMARY:
The aim of this study is to investigate the placental inflammation in women with gestational diabetes mellitus, in particular the role of inflammasome NLRP3 and the chemokine scavenger decoy receptor D6

DETAILED DESCRIPTION:
The aim of this study is to investigate systemic and placental inflammation in women with gestational diabetes mellitus, in particular the role of inflammasome NLRP3 and the chemokine scavenger decoy receptor D6, compared to women with uncomplicated pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Women with gestational diabetes mellitus
* Women with uncomplicated pregnancy
* Age >18 years
* Singleton pregnancy

Exclusion Criteria:

* Age < 18 years
* Infections (HIV,HCV)
* Multiple pregnancy
* Cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Placental inflammation | At delivery/birth
  Analysis of protein expression of inflammasome NLRP3 and D6 scavenger receptor in placental tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Tersigni, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy